CLINICAL TRIAL: NCT06352554
Title: Susceptibility Testing In Neisseria Gonorrhoeae (STING) Study
Brief Title: Susceptibility Testing In Neisseria Gonorrhoeae (STING) Study, Assessing the Performance of a New Rapid Test for Gonorrhoea Antibiotic Resistance, in a Cohort of 100 Culture Positive Neisseria Gonorrhoeae Infections
Acronym: STING
Status: Not yet recruiting | Type: Observational
Sponsor: SpeeDx Pty Ltd (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other); German Federal Ministry of Education and Research (Other Government); Australian Research Council Research Hub to Combat Antimicrobial Resistance (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023/ETH02474:STING; 224842/Z/21/Z (Other Grant/Funding Number: Wellcome Trust); 75A50122C00028 (Other Grant/Funding Number: HHS/BARDA OTA)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Diagnosis; Gonorrhea; Resistance Bacterial
MeSH Terms: conditions — Disease; Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to validate a novel antibiotic susceptibility test (InSignia) for gonorrhoea in patient clinical samples.

The hypothesis is that the InSignia test will be able to detect transcriptional responses after incubation in antibiotic for susceptible strains and not resistant strains.

Furthermore, this study will also add to our understanding on the performance of this test in various clinical specimens.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed/suspected NG infection
* Willingness to give written informed consent as well as to participate in and comply with the study.

Exclusion Criteria:

* Currently taking or having taken any antibiotics in the preceding 14 days
* English fluency below level required to understand study procedures
* Unwilling or unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting with confirmed NG infections in one or both of the following anatomical sites: the urethra & the rectum.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of performing antibiotic susceptibility testing (AST) for Neisseria gonorrhoeae directly from patient samples using InSignia workflow and assay against commonly used & clinically relevant antibiotics. | 1 year
  Feasibility of using the InSignia assay to determine the antibiotic susceptibility of NG - from sample collection, handling & transport to laboratory analysis & data interpretation.

SECONDARY OUTCOMES:
To study the performance of the InSignia assay in determining antibiotic susceptibility of NG against commonly used & clinically relevant agents in clinical samples with comparison to gold standard methods. | 1 year
  NG antibiotic susceptibility profile as determined by the InSignia assay compared to two other methods of NG AST - conventional culture via disc diffusion testing & E-test and genetic resistance testing via the ResistancePlus® GC (RPGC) IVD test (TGA, CE-IVD (IVDR) approved), developed by SpeeDx Pty Ltd.